CLINICAL TRIAL: NCT03042780
Title: Phase II Trial of FOLFIRINOX in Metastatic High Grade Gastroenteropancreatic Neuroendocrine Carcinomas
Brief Title: FOLFIRINOX in Metastatic High Grade Gastroenteropancreatic Neuroendocrine Carcinomas
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-18675
Record Dates: First submitted 2017-02-02; First posted 2017-02-03 (Estimated); Results first posted 2018-12-11 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Gastro-enteropancreatic Neuroendocrine Tumor; Pancreatic Cancer; Neuroendocrine Carcinomas of Pancreas; Islet Cell Carcinoma
Keywords: Gastroenteropancreatic neuroendocrine carcinomas (GEP-NECs); Metastatic; High grade; Pancreas; Neuroendocrine carcinoma of gastrointestinal tract
MeSH Terms: conditions — Gastro-enteropancreatic neuroendocrine tumor; Pancreatic Neoplasms; Carcinoma, Islet Cell; Neoplasm Metastasis | interventions — folfirinox; Granulocyte Colony-Stimulating Factor; Filgrastim; Cytokines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- FOLFIRINOX Treatment (Experimental): Participants will receive modified FOLFIRINOX which consists of 85 mg/m^2 of oxaliplatin, 400 mg/m^2 of leucovorin over the first 2 hours, 165 mg/m^2 of irinotecan in a 90-minute infusion on day 1, followed by a continuous, 46-hour infusion of 5-FU at a dosage of 2,400 mg/m^2. A cycle will be repeated every 14 days. Granulocyte colony-stimulating factor (G-CSF) prophylaxis will be allowed after each cycle. Participants will undergo re-staging studies every 8 weeks. Participants will receive up to 12 cycles during the study. Additional cycles will be determined per investigators' discretion.
  Interventions: Drug: FOLFIRINOX; Drug: Granulocyte colony-stimulating factor (G-CSF)

INTERVENTIONS:
Drug: FOLFIRINOX — The FOLFIRINOX regimen consists of oxaliplatin given as a 2-hour intravenous infusion, immediately followed by leucovorin given as a 2-hour intra-venous infusion, with the addition, after 30 minutes, of irinotecan given as a 90-minute intravenous infusion. This study treatment is immediately followed by a continuous intravenous infusion of 5-Fluorouracil (5-FU) over a 46-hour period every 2 weeks.
Drug: Granulocyte colony-stimulating factor (G-CSF) — The use of G-CSF will not be mandatory as primary prophylaxis, but will be allowed at investigators' discretion. If febrile neutropenia occurs, than the use of G-CSF will be mandatory after each following cycle of treatment.
  Other Names: Filgrastim; Cytokine

SUMMARY:
The purpose of this study is evaluate the efficacy and safety of FOLFIRINOX in patients with gastroenteropancreatic high-grade neuroendocrine carcinomas.

This is a prospective Phase II open-label trial, stratifying gastroenteropancreatic high grade neuroendocrine carcinomas participants equally into two cohorts (first-line versus beyond first-line).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed neuroendocrine carcinoma of the gastrointestinal (GI) tract. Potential participants with unknown origin for the neuroendocrine carcinoma in which a gastroenteropancreatic origin is suspected (per pathologist or investigator discretion) will be eligible for the study.
* Tumors must have a Ki-67 index greater than 20% and/or >20 mitotic figures/10 high-power fields.
* Must have metastatic disease.
* Must measurable disease, as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
* Any line of treatment (first line versus beyond first line).
* Age >18 years.
* Life expectancy of greater than 12 weeks.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.
* Must have adequate organ and marrow function.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Have had chemotherapy or radiotherapy within 3 weeks prior to entering the study.
* Receiving any other investigational agents.
* Untreated brain or meningeal metastases.
* Prior treatment with 5-fluorouracil (5-FU), irinotecan or oxaliplatin.
* Pre-treatment peripheral neuropathy greater than grade 1 per the CTCAE, version 4.0.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* A secondary primary cancer (excluding baso/squamous cell carcinoma of skin) within 1 year.
* Active viral hepatitis or autoimmune hepatitis. The work-up to confirm active hepatitis or autoimmune hepatitis will only be done if clinical suspicion based on investigator discretion.
* Potential participants with childbearing potential who are not willing to use adequate contraception precautions during the study and for 3 months after stopping study chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-01-03 (Actual); Study Completion 2018-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Strosberg, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- FOLFIRINOX Treatment: Participants will receive modified FOLFIRINOX which consists of 85 mg/m^2 of oxaliplatin, 400 mg/m^2 of leucovorin over the first 2 hours, 165 mg/m^2 of irinotecan in a 90-minute infusion on day 1, followed by a continuous, 46-hour infusion of 5-FU at a dosage of 2,400 mg/m^2. A cycle will be repeated every 14 days. Granulocyte colony-stimulating factor (G-CSF) prophylaxis will be allowed after each cycle. Participants will undergo re-staging studies every 8 weeks. Participants will receive up to 12 cycles during the study. Additional cycles will be determined per investigators' discretion.
  FOLFIRINOX: The FOLFIRINOX regimen consists of oxaliplatin given as a 2-hour intravenous infusion, immediately followed by leucovorin given as a 2-hour intra-venous infusion, with the addition, after 30 minutes, of irinotecan given as a 90-minute intravenous infusion. This study treatment is immediately followed by a continuous intravenous infusion of 5-Fluorouracil (5-FU) over a 46-hour period
Period: Overall Study
Arm/Group | FOLFIRINOX Treatment
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- FOLFIRINOX Treatment: Participants will receive modified FOLFIRINOX which consists of 85 mg/m^2 of oxaliplatin, 400 mg/m^2 of leucovorin over the first 2 hours, 165 mg/m^2 of irinotecan in a 90-minute infusion on day 1, followed by a continuous, 46-hour infusion of 5-FU at a dosage of 2,400 mg/m^2. A cycle will be repeated every 14 days. Participants will receive up to 12 cycles during the study. Additional cycles will be determined per investigators' discretion.
Arm/Group | FOLFIRINOX Treatment
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Radiographic Response Rate (ORR)
Description: The primary efficacy endpoint is objective response rate as determined by radiology review, as defined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Complete Response (CR): complete disappearance of all target lesions. Partial Response (PR): at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum longest diameter. Progressive disease (PD): at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this may include the baseline sum). Stable Disease (SD): neither sufficient decrease to qualify for partial response nor sufficient increase to qualify for progressive disease.
Time Frame: Up to 36 months
Population: Due to low accrual, study was halted prematurely. No data, as no patients were analyzed.
Arm/Group | FOLFIRINOX Treatment
Number analyzed (Participants) | 0

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS: from initiation date of therapy to disease progression or death. Progressive disease (PD): at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this may include the baseline sum).
Time Frame: Up to 36 months
Population: No data displayed because Outcome Measure has zero total participants analyzed.
Arm/Group | FOLFIRINOX Treatment
Number analyzed (Participants) | 0

3. Other Pre Specified Outcome: Treatment Related Morbidity
Description: Safety analysis will be analyzed by collecting date on treatment-related morbidity and mortality. Investigators will collect data on frequency, type and severity of all adverse events that occur on or after Cycle 1, Day 1 according to National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE; Version 4.0).
Time Frame: Up to 36 months
Population: No data displayed because Outcome Measure has zero total participants analyzed.
Arm/Group | FOLFIRINOX Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- FOLFIRINOX Treatment: Participants received modified FOLFIRINOX which consists of 85 mg/m^2 of oxaliplatin, 400 mg/m^2 of leucovorin over the first 2 hours, 165 mg/m^2 of irinotecan in a 90-minute infusion on day 1, followed by a continuous, 46-hour infusion of 5-FU at a dosage of 2,400 mg/m^2. A cycle will be repeated every 14 days. Granulocyte colony-stimulating factor (G-CSF) prophylaxis will be allowed after each cycle.
Arm/Group | FOLFIRINOX Treatment
All-Cause Mortality (participants affected / at risk) | 1/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOLFIRINOX Treatment (N=2)
Anemia (Blood and lymphatic system disorders) | 1 (4)
Blurred Vision (Eye disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Skin Infection (Infections and infestations) | 1 (1) — right forearm ant bite
Alanine aminotransferase increased (Investigations) | 1 (7)
Alkaline phosphatase increased (Investigations) | 1 (4)
Aspartate aminotransferase increased (Investigations) | 1 (6)
Lymphocyte count decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (3)
White blood cell decreased (Investigations) | 2 (5)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) — Body aches, joint pain
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study terminated early due to inability to accrue, leading to small number of participants analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-14): https://cdn.clinicaltrials.gov/large-docs/80/NCT03042780/Prot_SAP_000.pdf